CLINICAL TRIAL: NCT00403754
Title: A Randomized, Double-blind, Placebo-controlled, 4-period 4-treatment Crossover, Multicenter, Single-dose, Dose-ranging Study Followed by a Single Day's Treatment With Open Label Salmeterol Bid (100 µg/Day), to Assess the Efficacy and Safety of 3 Doses of Indacaterol (150, 300, & 600 µg) Delivered Via Single Dose Dry Powder Inhaler (SDDPI) in Japanese Asthma Patients
Brief Title: Dose Ranging Study for Indacaterol in Japanese Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149A1202
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Asthma
Keywords: asthma; QAB149; indacaterol; long acting β2-agonist; bronchodilator
MeSH Terms: conditions — Asthma | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo-Ind 150 μg-Ind 300 μg-Ind 600 μg-Salmeterol (Experimental): In treatment period 1: patients received 2 placebo capsules; in treatment period 2: patients received 1 indacaterol (Ind) 150 μg capsule + 1 placebo capsule; in treatment period 3: patients received 1 indacaterol 300 μg capsule + 1 placebo capsule; and in treatment period 4: patients received 2 indacaterol 300 μg capsules. Two inhalation capsules of study drug were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of each treatment period at approximately the same time of day +/- 15 minutes. There was a washout period of 14-28 days between each treatment period. In open label treatment period 5: patients received 100 μg salmeterol (50 μg in the morning, 50 μg twelve hours post initial dose) inhaled via Diskus®, an inhalation device, on Day 1.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Ind 150 μg-Ind 600 μg-Placebo-Ind 300 μg-Salmeterol (Experimental): In treatment period 1: patients received 1 indacaterol (Ind) 150 μg capsule + 1 placebo capsule; in treatment period 2: patients received 2 indacaterol 300 μg capsules; in treatment period 3: patients received 2 placebo capsules; and in treatment period 4: patients received 1 indacaterol 300 μg capsule + 1 placebo capsule. Two inhalation capsules of study drug were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of each treatment period at approximately the same time of day +/- 15 minutes. There was a washout period of 14-28 days between each treatment period. In open label treatment period 5: patients received 100 μg salmeterol (50 μg in the morning, 50 μg twelve hours post initial dose) inhaled via Diskus®, an inhalation device, on Day 1.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol (Experimental): In treatment period 1: patients received 1 indacaterol (Ind) 300 μg capsule + 1 placebo capsule; in treatment period 2: patients received 2 placebo capsules; in treatment period 3: patients received 2 indacaterol 300 μg capsules; and in treatment period 4: patients received 1 indacaterol 150 μg capsule + 1 placebo capsule. Two inhalation capsules of study drug were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of each treatment period at approximately the same time of day +/- 15 minutes. There was a washout period of 14-28 days between each treatment period. In open label treatment period 5: patients received 100 μg salmeterol (50 μg in the morning, 50 μg twelve hours post initial dose) inhaled via Diskus®, an inhalation, device on Day 1.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Ind 600 μg-Ind 300 μg-Ind 150 μg-Placebo-Salmeterol (Experimental): In treatment period 1: patients received 2 indacaterol (Ind) 300 μg capsules; in treatment period 2: patients received 1 indacaterol 300 μg capsule + 1 placebo capsule; in treatment period 3: patients received 1 indacaterol 150 μg capsule + 1 placebo capsule; and in treatment period 4: patients received 2 placebo capsules. Two inhalation capsules of study drug were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of each treatment period at approximately the same time of day +/- 15 minutes. There was a washout period of 14-28 days between each treatment period. In open label treatment period 5: patients received 100 μg salmeterol (50 μg in the morning, 50 μg twelve hours post initial dose) inhaled via Diskus®, an inhalation device, on Day 1.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol

INTERVENTIONS:
Drug: Indacaterol — In the morning, powder filled capsules inhaled using a single dose dry powder inhaler (SDDPI).
  Other Names: QAB149
Drug: Placebo — Placebo to indacaterol was provided in powder filled capsules with a single dose dry powder inhaler (SDDPI).
Drug: Salmeterol — Salmeterol 100 μg total dose taken on Day 1. 50 μg in the morning and 50 μg twelve hours post initial dose inhaled via Diskus®, an inhalation device for Salmeterol.
  Other Names: Serevent

SUMMARY:
This study was designed to provide data about the safety and efficacy of 3 doses of indacaterol (150, 300, and 600 µg) in Japanese asthma patients so that an optimal dose, or doses, could be chosen for testing in later studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Japanese asthmatic patients aged 18 to 75 years old.

Exclusion Criteria:

* Patients who have been hospitalized or had emergency room treatment for an acute asthma attack in the 6 months prior to the first day of screening or during the screening period.
* Patients who have used tobacco products within 6 months prior to the first day of screening or have a smoking history of greater than 10 pack years.
* Patients with a history of malignancy with the exception of localized basal cell carcinoma of the skin.
* Pregnant or nursing (lactating) women.
* Patients who have had treatment with disallowed medications including investigational drug.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Principal Investigator — Novartis Pharmaceuticals Japan
Locations (8):
- Japan (8):
  - Novartis Investigative Site, Kasukabe
  - Novartis Investigator Site, Kishiwada
  - Novartis Investigative Site, Shimotsuga
  - Novartis Investigator Site, Suita
  - Novartis Investigative Site, Tokyo
  - Novartis, Tokyo
  - Novartis Investigator Site, Wakayama
  - Novartis Investigator Site, Yokohama

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 14 day eligibility screening period insured all participants were stable on their permissible asthma treatment before proceeding onto core study drug treatment.
Groups:
- Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol: In treatment period 1: patients received 1 indacaterol (Ind) 300 μg capsule + 1 placebo capsule; in treatment period 2: patients received 2 placebo capsules; in treatment period 3: patients received 2 indacaterol 300 μg capsules; and in treatment period 4: patients received 1 indacaterol 150 μg capsule + 1 placebo capsule. Two inhalation capsules of study drug were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of each treatment period at approximately the same time of day +/- 15 minutes. There was a washout period of 14-28 days between each treatment period. In open label treatment period 5: patients received 100 μg salmeterol (50 μg in the morning, 50 μg twelve hours post initial dose) inhaled via Diskus®, an inhalation, device on Day 1.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use t
- Ind 600 μg-Ind 300 μg-Ind150 μg-Placebo-Salmeterol: In treatment period 1: patients received 2 indacaterol (Ind) 300 μg capsules; in treatment period 2: patients received 1 indacaterol 300 μg capsule + 1 placebo capsule; in treatment period 3: patients received 1 indacaterol 150 μg capsule + 1 placebo capsule; and in treatment period 4: patients received 2 placebo capsules. Two inhalation capsules of study drug were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of each treatment period at approximately the same time of day +/- 15 minutes. There was a washout period of 14-28 days between each treatment period. In open label treatment period 5: patients received 100 μg salmeterol (50 μg in the morning, 50 μg twelve hours post initial dose) inhaled via Diskus®, an inhalation device, on Day 1.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use t
Period: Core Treatment Period 1
Arm/Group | Placebo-Ind 150 μg-Ind 300 μg-Ind 600 μg-Salmeterol | Ind 150 μg-Ind 600 μg-Placebo-Ind 300 μg-Salmeterol | Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol | Ind 600 μg-Ind 300 μg-Ind150 μg-Placebo-Salmeterol
Started | 11 | 10 | 9 | 11
Completed | 11 | 9 | 9 | 11
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Core Treatment Period 2
Arm/Group | Placebo-Ind 150 μg-Ind 300 μg-Ind 600 μg-Salmeterol | Ind 150 μg-Ind 600 μg-Placebo-Ind 300 μg-Salmeterol | Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol | Ind 600 μg-Ind 300 μg-Ind150 μg-Placebo-Salmeterol
Started | 11 | 9 | 9 | 11
Completed | 11 | 9 | 8 | 11
Not Completed | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Period: Core Treatment Period 3
Arm/Group | Placebo-Ind 150 μg-Ind 300 μg-Ind 600 μg-Salmeterol | Ind 150 μg-Ind 600 μg-Placebo-Ind 300 μg-Salmeterol | Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol | Ind 600 μg-Ind 300 μg-Ind150 μg-Placebo-Salmeterol
Started | 11 | 9 | 8 | 11
Completed | 11 | 9 | 8 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Core Treatment Period 4
Arm/Group | Placebo-Ind 150 μg-Ind 300 μg-Ind 600 μg-Salmeterol | Ind 150 μg-Ind 600 μg-Placebo-Ind 300 μg-Salmeterol | Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol | Ind 600 μg-Ind 300 μg-Ind150 μg-Placebo-Salmeterol
Started | 11 | 9 | 8 | 11
Completed | 11 | 9 | 8 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Open Label: Salmeterol
Arm/Group | Placebo-Ind 150 μg-Ind 300 μg-Ind 600 μg-Salmeterol | Ind 150 μg-Ind 600 μg-Placebo-Ind 300 μg-Salmeterol | Ind 300 μg-Placebo-Ind 600 μg-Ind 150 μg-Salmeterol | Ind 600 μg-Ind 300 μg-Ind150 μg-Placebo-Salmeterol
Started | 11 | 9 | 8 | 11
Completed | 11 | 9 | 8 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population included all 4 treatment groups who received indacaterol 150 µg, 300 µg, and 600 µg and placebo via a single dose dry powder inhaler (SDDPI) in the 4 different sequences of the core phase. Two capsules of study medication were inhaled in the morning on Day 1 of each treatment period. Following the core phase patients continued to the Salmeterol open label phase. Salmeterol was inhaled via a Diskus inhalation device 50 µg in the morning and 50 µg 12 hours post initial dose on Day 1. Patients received each treatment only once.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 22 to 24 Hours Post-dose on Day 2
Description: Spirometry was conducted according to internationally accepted standards. Standardized area under the curve (AUC22-24h) of FEV1 values taken at 22, 23 and 24 hours post dose, was calculated based on the trapezoidal rule. Analysis of Covariance was carried out with a mixed model that used (period) baseline, defined as the value of FEV1 measured prior to the first study drug intake in the period, as a covariate.
Time Frame: 22, 23, and 24 hours post-dose on Day 2
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol 600 µg: Two capsules of indacaterol 300 µg were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning on Day 1 of the treatment period. Indacaterol 600 µg was administered only once to each patient.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Indacaterol 300 µg: One capsule of indacaterol 300 µg and 1 placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning on Day 1 of the treatment period. Indacaterol 300 µg was administered only once to each patient.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Indacaterol 150 µg: One capsule of indacaterol 150 µg and 1 placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning on Day 1 of the treatment period. Indacaterol 150 µg was administered only once to each patient.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Placebo: Two placebo capsules were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning on Day 1 of the treatment period. Placebo was administered to each patient only once.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Salmeterol 100 μg: Open label Salmeterol 100 μg total dose taken on Day 1. 50 μg in the morning and 50 μg twelve hours post initial dose inhaled via Diskus®, an inhalation device for Salmeterol.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 600 µg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo | Salmeterol 100 μg
Number analyzed (Participants) | 39 | 40 | 40 | 40 | 39
Liters | 2.31 (0.023) | 2.28 (0.022) | 2.24 (0.022) | 2.06 (0.022) | 2.23 (0.022)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) by Time Point From 5 Minutes to 12 Hours Post-dose on Day 1 and From 22 to 24 Hours Post-dose on Day 2
Description: Spirometry was conducted according to internationally accepted standards. FEV1 by time point was calculated using a mixed model with (period) baseline, defined as the value measured prior to the first study drug intake in the period, as a covariate.
Time Frame: 5, 15, and 30 minutes; and 1, 2, 4, 8, and 12 hours post-dose on Day 1; and 22, 23, and 24 hours post-dose on Day 2
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 600 µg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo | Salmeterol 100 μg
Number analyzed (Participants) | 39 | 40 | 40 | 40 | 39
Liters
  5 minutes | 2.25 [2.22 to 2.27] | 2.20 [2.18 to 2.23] | 2.19 [2.16 to 2.22] | 2.04 [2.01 to 2.07] | 2.13 [2.10 to 2.15]
  15 minutes | 2.33 [2.30 to 2.36] | 2.28 [2.25 to 2.32] | 2.27 [2.24 to 2.30] | 2.05 [2.02 to 2.08] | 2.19 [2.16 to 2.22]
  30 minutes | 2.37 [2.34 to 2.41] | 2.33 [2.30 to 2.37] | 2.30 [2.27 to 2.34] | 2.07 [2.03 to 2.10] | 2.24 [2.21 to 2.27]
  1 hour | 2.41 [2.38 to 2.45] | 2.35 [2.32 to 2.38] | 2.32 [2.29 to 2.35] | 2.09 [2.06 to 2.12] | 2.29 [2.25 to 2.32]
  2 hours | 2.45 [2.41 to 2.48] | 2.39 [2.35 to 2.43] | 2.38 [2.34 to 2.42] | 2.13 [2.09 to 2.16] | 2.34 [2.30 to 2.37]
  4 hours | 2.42 [2.38 to 2.47] | 2.39 [2.35 to 2.43] | 2.35 [2.31 to 2.39] | 2.10 [2.06 to 2.14] | 2.34 [2.30 to 2.38]
  8 hours | 2.37 [2.33 to 2.41] | 2.35 [2.31 to 2.38] | 2.28 [2.24 to 2.31] | 2.06 [2.02 to 2.09] | 2.25 [2.21 to 2.29]
  12 hours | 2.33 [2.28 to 2.37] | 2.30 [2.26 to 2.34] | 2.24 [2.20 to 2.28] | 2.00 [1.96 to 2.05] | 2.20 [2.16 to 2.24]
  22 hours | 2.30 [2.26 to 2.34] | 2.25 [2.21 to 2.29] | 2.20 [2.16 to 2.24] | 2.01 [1.97 to 2.05] | 2.18 [2.14 to 2.22]
  23 hours | 2.32 [2.28 to 2.36] | 2.28 [2.25 to 2.32] | 2.25 [2.21 to 2.29] | 2.06 [2.02 to 2.10] | 2.23 [2.20 to 2.27]
  24 hours | 2.32 [2.28 to 2.35] | 2.29 [2.25 to 2.33] | 2.26 [2.22 to 2.30] | 2.09 [2.06 to 2.13] | 2.27 [2.23 to 2.31]

3. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) From 5 Minutes to 4 Hours Post-dose on Day 1
Description: Spirometry was conducted according to internationally accepted standards. Peak FEV1 is the maximum FEV1 recorded in the period between 5 minutes and 4 hours post dose. Analysis of Covariance was carried out with a mixed model that used (period) baseline, defined as the value of FEV1 measured prior to the first study drug intake in the period, as a covariate.
Time Frame: 5 minutes to 4 hours post-dose on Day 1
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 600 µg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo | Salmeterol 100 μg
Number analyzed (Participants) | 39 | 40 | 40 | 40 | 39
Liters | 2.49 (0.018) | 2.44 (0.018) | 2.41 (0.018) | 2.19 (0.18) | 2.39 (0.018)

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 5 Minutes Post-dose on Day 1 to 24 Hours Post-dose on Day 2
Description: Spirometry was conducted according to internationally accepted standards. Standardized area under the curve (AUC0-24h) of FEV1 values taken at pre-dose to 24 hours post dose was calculated based on the trapezoidal rule. Analysis of Covariance was carried out with a mixed model that used (period) baseline, defined as the value of FEV1 measured prior to the first study drug intake in the period, as a covariate.
Time Frame: 5 minutes to 12 hours post-dose on Day 1; and 22 to 24 hours post-dose on Day 2
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 600 µg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo | Salmeterol 100 μg
Number analyzed (Participants) | 39 | 40 | 40 | 40 | 39
Liters | 2.35 (0.022) | 2.31 (0.021) | 2.26 (0.021) | 2.04 (0.021) | 2.24 (0.021)

ADVERSE EVENTS:
Description: Safety Population included all participants who received at least one dose of study drug.
Groups:
- Indacaterol 150 μg: 1 Indacaterol 150 μg capsule + 1 Placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of the Indacaterol 150 μg treatment period.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Indacaterol 300 μg: 1 Indacaterol 300 μg capsules + 1 Placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of the Indacaterol 300 μg treatment period.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Indacaterol 600 μg: 2 Indacaterol 300 μg capsules were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of the Indacaterol 600 μg treatment period.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
- Placebo: 2 Placebo capsules were inhaled using a single dose dry powder inhaler (SDDPI) in the morning on day 1 of the Placebo treatment period.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Indacaterol 600 μg | Placebo | Salmeterol 100 μg
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/39 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 14/40 | 14/40 | 14/39 | 6/40 | 1/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=40) | Indacaterol 300 μg (N=40) | Indacaterol 600 μg (N=39) | Placebo (N=40) | Salmeterol 100 μg (N=39)
HEADACHE (Nervous system disorders) | 2 | 2 | 1 | 3 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 | 13 | 14 | 3 | 0
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.